CLINICAL TRIAL: NCT05181540
Title: A Phase 3 Double-Blind, Randomized, Placebo Controlled Study to Evaluate the Efficacy and Safety of AB-205 Plus Standard of Care Versus Placebo Plus Standard of Care in Adults With Lymphoma Undergoing High-Dose Therapy and Autologous Hematopoietic Cell Transplantation (HDT-AHCT) (E-CELERATE)
Brief Title: A Study of the Effects of AB-205 in Patients With Lymphoma Undergoing Autologous Hematopoietic Cell Transplantation
Acronym: E-CELERATE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Interim analysis showed lack of efficacy
Sponsor: Angiocrine Bioscience (Industry)
Collaborators: California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: AB-205-301
Record Dates: First submitted 2021-12-16; First posted 2022-01-06 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Hodgkin Lymphoma; Non Hodgkin Lymphoma
Keywords: Lymphoma; Cellular Therapy
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin; Lymphoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AB-205 plus standard-of-care preventive and supportive therapies. (Experimental)
  Interventions: Biological: AB-205
- Placebo plus standard-of-care preventive and supportive therapies. (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: AB-205 — Allogeneic genetically engineered human umbilical vein endothelial cells
  Other Names: E-CEL cells
  Arms: AB-205 plus standard-of-care preventive and supportive therapies.
Other: Placebo — Placebo
  Arms: Placebo plus standard-of-care preventive and supportive therapies.

SUMMARY:
High-dose chemotherapy followed by blood stem cell transplantation is administered to lymphoma patients with an intention to cure. However, high-dose chemotherapy simultaneously causes damage to healthy tissues that frequently result in severe complications that lead to hospitalization and can be life threatening. These severe complications involve the blood, immune, gastro-intestinal systems, and other vital organs.

The purpose of this study is to determine if experimental therapy AB-205 (study drug) can prevent or reduce the occurrence and duration of the severe chemotherapy related complications when compared to placebo in patients with lymphoma undergoing treatment with high-dose chemotherapy and blood stem cell transplantation. All patients, whether treated with AB-205 or placebo, will receive standard preventive and supportive care therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 40 years old
2. Diagnosis of Hodgkin lymphoma (HL) or non-Hodgkin lymphoma (NHL)
3. Candidates for HDT-AHCT with one of the following conditioning regimens:

   1. BEAM (carmustine, etoposide, cytarabine, melphalan)
   2. BeEAM (bendamustine, etoposide, cytarabine, melphalan)
4. Achieved CR or PR prior to planned HDT
5. ECOG ≤ 2
6. Weight ≤ 1.6 × ideal body weight (IBW) per Devine formula
7. Serum bilirubin ≤ 2 mg/dL, unless benign congenital hyperbilirubinemia
8. AST, ALT, and alkaline phosphatase < 3 × ULN
9. Creatinine clearance ≥ 30 ml/min (calculated by Cockcroft Gault)
10. LVEF ≥ 45% by MUGA or resting echocardiogram
11. Pulmonary function (FEV1 and corrected DLCO) ≥ 45% predicted
12. Willingness and ability to comply with scheduled visits, drug administration plan, protocol-specified laboratory tests, other study procedures, and study restrictions
13. Sexually active females of childbearing potential must have a negative urine pregnancy test and agree to use two accepted methods of contraception during the study and for 3 months after their last dose of study drug.
14. Male subjects who are sexually active and who are partners of females of childbearing potential: agreement to use two forms of contraception as in criterion 12 above and to not donate sperm during the treatment period and for at least 3 months after the last dose of study drug
15. Ability to provide written informed consent.

Exclusion Criteria:

1. History of prior HCT
2. Primary CNS lymphoma
3. Lymphoma with CNS involvement at time of relapse prior to planned HDT-AHCT
4. Active malignancy other than the one for which the subject is undergoing HDT AHCT. Subjects with cervical carcinoma in situ or localized basal or squamous cell carcinoma treated with definitive surgery are eligible
5. Subjects with a serious concomitant medical condition that could interfere with the conduct of the clinical trial, such as unstable angina, renal failure requiring hemodialysis, or active infection requiring IV antibiotics
6. Subjects with a known history of HIV
7. Subjects who have known hypersensitivity reactions to bovine (cow) proteins or documented allergy to DMSO
8. Subject has other conditions that in the opinion of the investigator would require reduced dose (intensity) of BEAM or BeEAM regimens

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
The absence of oral/GI severe regimen related toxicities (oral/GI SRRT). | 21 Days

SECONDARY OUTCOMES:
Duration of oral/GI SRRT | 21 Days
Symptom burden per MD Anderson Symptom Inventory (MDASI) | 21 Days
Duration of febrile neutropenia | 21 Days
Time to neutrophil engraftment | 21 Days

CONTACTS AND LOCATIONS:
Overall Officials: Paul Finnegan, MD, Study Director — Angiocrine Bioscience, Inc.
Locations (28):
- United States (28):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - University of California, Los Angeles, Los Angeles, California
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - UC San Diego Moores Cancer Center, San Diego, California
  - Sarah Cannon Research Institute, Colorado, Denver, Colorado
  - Medstar Georgetown University Hospital, Washington D.C., District of Columbia
  - University of Miami - Sylvester Comprehensive Cancer Center, Miami, Florida
  - University of South Florida (USF) - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University - Winship Cancer Institute, Atlanta, Georgia
  - University of Illinois Cancer Center, Chicago, Illinois
  - Indiana University Simon Comprehensive Cancer Center, Indianapolis, Indiana
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - University Of Maryland School Of Medicine, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota Medical Center, Fairview, Minneapolis, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medical College/New York Presbyterian Hospital, New York, New York
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No